CLINICAL TRIAL: NCT03924479
Title: Respiratory Muscle-mediated Neural and Cardiovascular Consequences in Heart Failure With Preserved Ejection Fraction
Brief Title: Respiratory Muscle Function in Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Thomas P. Olson, M.S., Ph.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 17-007785
Record Dates: First submitted 2019-02-04; First posted 2019-04-23 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure, Diastolic
Keywords: heart failure preserved ejection fraction; exercise; respiratory muscle
MeSH Terms: conditions — Heart Failure, Diastolic; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing muscle training (Experimental): The breathing muscle training will consist of 7 sessions per week (1 per day) for 8 weeks. Each training session will consist of breathing ~15 times each minute for 30 minutes at 40% of maximal breathing muscle strength, while using the breathing muscle trainer. During the inhalation, participants will be instructed to inhale as fast as they can, while exhalations will be performed at the participants discretion.
  Interventions: Device: PowerBreathe (Breathing muscle training)
- Sham breathing muscle training (Sham Comparator): The breathing muscle training will consist of 7 sessions per week (1 per day) for 8 weeks. Each training session will consist of breathing ~15 times each minute for 30 minutes at 2%% of maximal breathing muscle strength, while using the breathing muscle trainer. During the inhalation, participants will be instructed to inhale as fast as they can, while exhalations will be performed at the participants discretion.
  Interventions: Device: PowerBreathe (Breathing muscle training)

INTERVENTIONS:
Device: PowerBreathe (Breathing muscle training) — The breathing muscle breathing training will consist of using the PowerBreathe training for 8 weeks. The PowerBreathe is an inspiratory pressure threshold trainer.The valve blocks the airflow until the threshold pressure is achieved by breathing in forcefully into the device.
  Other Names: PowerBreathe Device

SUMMARY:
This study is being done because investigators are trying to determine how respiratory muscle and lung function influence the exercise responses in heart failure and healthy participants. Further, the heart failure patients will participate in an intervention to improve their respiratory muscle function to determine if this improves exercise capacity.

DETAILED DESCRIPTION:
The participants enrolled in this study will be asked to make 4 or 9 separate study visits. Healthy participants will perform 4 study visits and heart failure participants will perform 9 study visits.

During study visit 1, the participants will be asked to get a DEXA bone scan, perform pulmonary function tests, and exercise on a stationary bike at maximal exertion while breathing into a mouth piece. During the exercise test, a iodine-based dye will be injected via a venous catheter in the arm. Also, a thin balloon will be inserted through the nose into the esophagus.

During study visit 2, the participants will breathe the same way they did during exercise, but will be seated and not exercising. A thin balloon will be inserted through the nose into the esophagus.

During study visits 3 and 4, the participants will perform different respiratory muscle workouts at rest that will be at different intensities ranging from very easy to moderate for ~10 minutes. An iodine-based dye will be injected via a venous catheter in the arm.

The participant's with heart failure will then perform 8 weeks of breathing muscle training at home. After 3 weeks of breathing muscle training, the participants will return for study visit 5 where the training load will be adjusted. Following the 8 weeks of breathing muscle training, the heart failure participants will perform the same 4 study visits as outlined above.

ELIGIBILITY:
Healthy subjects: Adults (≥21 years of age) in the absence of a history of HFpEF or HFrEF, pulmonary, neurologic, orthopedic, or other diseases affecting the neuromuscular system. Controls will be matched for age and sex.

All HFpEF patients will be managed by their primary care physician or cardiologist with additional review and oversight by Dr. Borlaug (Co-Investigator) prior to enrollment to ensure adequacy of inclusion and exclusion criteria and that participation in exercise testing and resistance exercise training is safe.

Inclusion Criteria for HFpEF, includes:

* Clinical diagnosis of HFpEF.
* Patients with a history stable (no medication changes in past 6 weeks (w/duration of diagnosis >6 months).
* New York Heart Association class I-III.
* Current non-smokers with <15 pack year history.
* Non-pregnant women, and individuals who are able to exercise (i.e. without orthopedic limitations or neuromuscular disorders).

Exclusion Criteria for all subjects, includes:

* history of dangerous arrhythmias
* body mass index >35 kg/m2
* current smokers and/or smoking history >15 pack years
* pregnant women
* uremia, history of allergy to iodides
* impaired renal function
* creatinine value greater than or equal to 1.3 mg/dL (via clinical record within the past 6 months)
* diagnosis of liver disease
* individuals who are not able to engage in exercise

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-21 (Actual)

PRIMARY OUTCOMES:
Breathing muscle oxygen cost | Year 1
  Breathing muscle oxygen uptake between heart failure and healthy participants
Respiratory muscle blood flow | Year 1
  Breathing muscle blood flow between heart failure and healthy participants
Systolic and diastolic blood pressure | Year 1
  Respiratory muscle workout-induced increases in systolic and diastolic blood pressure between heart failure and healthy participants
Breathing muscle oxygen cost | Year 2
  Breathing muscle oxygen uptake from pre to post-breathing muscle training in heart failure participants
Respiratory muscle blood flow | Year 2
  Breathing muscle blood flow rom pre to post-breathing muscle training in heart failure participants
Systolic and diastolic blood pressure | Year 2
  Respiratory muscle workout-induced increases in systolic and diastolic blood pressure from pre to post-breathing muscle training in heart failure participants

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P Olson, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials